CLINICAL TRIAL: NCT05648552
Title: Altered Structural-functional Connectivity Coupling on Chronic Subcortical Stroke: a Resting-state fMRI Study
Brief Title: Altered Structural-functional Connectivity Coupling on Chronic Subcortical Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-PY-27
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Motor Activity
Keywords: Stroke; Motor dysfunction; MRI; structural connectivity; functional connectivity
MeSH Terms: conditions — Stroke; Motor Activity; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke group: Chronic subcortical stroke participants with motor dysfunction
- Healthy controls group: Well-matched healthy controls

SUMMARY:
The current study aims to reveal the SC-FC coupling pattern and its relationship with motor function in post-stroke survivors with motor dysfunction by multimodal MRI.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and disability in China. Recently, many previous studies suggested exploring the functional reorganization of the motor function among post-stroke survivors is urgent to be solved in both clinical work and applied basic research. Investigating the structural connectivity (SC) of the brain could visualize the anatomical connections between different brain regions and exploring the functional connectivity (FC) could reveal the functional activity patterns of the human brain in resting- and task- states. Previous studies suggested that SC-FC coupling analysis may shed light on exploring biological markers for the assessment and treatment of motor deficits in post-stroke survivors. The current study aims to reveal the SC-FC coupling pattern and its relationship with motor function in post-stroke survivors with motor dysfunction by multimodal MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with the diagnostic criteria of "Stroke" in the 2010 "Guidelines for the Prevention and Treatment of Cerebrovascular Diseases in China," and confirmed by head CT or MRI.
2. First onset unilateral subcortical stroke (basal ganglia, thalamus, internal capsule, corona radiata, lateral ventricles, etc.).
3. Age ranged from 30 to 75 years old.
4. Right-handedness before stroke.
5. Greater than three months since stroke onset and Brunnstrom graded as III-VI; 6. The condition and vital signs are stable.

7. Sign the informed consent form.

Exclusion Criteria:

1. Any contraindications for the MRI examination.
2. History of other brain diseases and drug dependency.
3. Unstable conditions or accompanied by malignant and rapidly progressing diseases, such as severe atrial fibrillation.
4. Serious communication barriers, cognitive impairment, or cooperation with difficulties.

Ages: 30 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To recruit 35 chronic subcortical post-stroke participants with motor dysfunction and 35 well-matched healthy controls from the Department of Rehabilitation Medicine of Nanjing Drum Tower Hospital and the local communities.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Structural-functional Connectivity Coupling | Within 1 week after enrollment
  The coupling between structural connectivity and functional connectivity
Fugl-Meyer Assessment | Within 1 week after enrollment
  Assessing the motor function in post-stroke participants

SECONDARY OUTCOMES:
Chinese version of Modified Barthel Index | Within 1 week after enrollment
  Assessing the activities of daily living in post-stroke participants
Broetz Hand Test | Within 1 week after enrollment
  Assessing the hemiplegic hand performance in post-stroke participants
Placebo Questionnaire | Within 1 week after enrollment
  Self-evaluation of rehabilitation treatment in post-stroke participants
Hamilton Depression Rating Scale | Within 1 week after enrollment
  Assessing the depression in post-stroke participants
Chinese (Putonghua) Version of Oxford Cognitive Screen | Within 1 week after enrollment
  Assessing the cognition in post-stroke participants

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Hong, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong W, Liu Z, Zhang X, Li M, Yu Z, Wang Y, Wang M, Wu Y, Fang S, Yang B, Xu R, Zhao Z. Distance-related functional reorganization predicts motor outcome in stroke patients. BMC Med. 2024 Jun 18;22(1):247. doi: 10.1186/s12916-024-03435-7. PMID 38886774